CLINICAL TRIAL: NCT00198874
Title: Youth Drug Abuse Family and Cognitive-Behavioral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA010777-08 (NIH); 5R01DA010777-08 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Drug Abuse
Keywords: drug abuse; drug dependence; treatment; randomized trial; stage II study; adolescents; young adults; efficacy study
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy; Educational Status

ARMS (4):
- Psychoeducation (Active Comparator)
  Interventions: Other: Education
- Conitive Behavorial Therapy (Experimental)
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Therapy
- Family Therapy (Experimental)
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Therapy
- Intergrated Family (Experimental)
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Integrated Family and Cognitive-Behavioral Therapy — The family therapy component of IFCBT includes engagement, active treatment, and maintenance phases. The cognitive program focuses on harmful effects of drugs and strategies to better manage drug abuse risks. The cognitive-behavioral program introduces youths to problem-solving behavior change principles and study skills to promote school achievement.
  Arms: Conitive Behavorial Therapy; Family Therapy; Intergrated Family
Other: Education — Drug education curriculum was delivered to participants assigned to this condition.
  Arms: Psychoeducation

SUMMARY:
This Stage II study is in response to NIDA's Behavioral Therapies Development Program (PA-99-107). A randomized clinical trial is proposed to evaluate the direct, mediated, and moderated effects of Integrated Family and Cognitive-Behavioral Therapy (IFCBT), a multisystems treatment for adolescent drug abuse with promising efficacy results. In the first study aim, we seek to evaluate the separate and possibly synergistic effects of family systems and cognitive-behavioral IFCBT components on posttreatment drug abuse problem severity, problem behavior, psychiatric distress, and academic achievement of adolescent drug abusers. Innovative analytic strategies are subsequently used to evaluate the degree to which successful outcomes are attributable to specific familial and cognitive-behavioral change processes targeted by IFCBT components. The possibility of effect-modification also is considered, with a focus on neurocognitive, psychiatric comorbidity, and demographic factors. Namely, we seek to understand how variations in specific client characteristics, such as executive dysfunctions or psychiatric comorbidity, might explain why treatments work for some drug abusing youths but not others. In addition to promising findings on IFCBT efficacy, this Stage II proposal benefits from the development and Stage I study application of (a) treatment manuals; (b) therapist training procedures; (c) therapist adherence and competence tools; (d) a neuropsychological battery to assess cognitive functions; (e) a psychodiagnostic battery to assess comorbid psychiatric disorders; and (f) a study assessment battery comprised of therapeutic process and outcome measures. This revised application has sought to address well-taken concerns cited by the reviewers while maintaining proposal strengths. The lack of adolescent drug treatment research continues to be a serious gap in the addictions literature despite alarmingly high rates of drug abuse among youth and the range of morbidities and mortality that result nationwide. If successful, this project should help to identify specific behavior change processes targeted by family systems and cognitive-behavioral treatments that foster subsequent reductions in drug use and problem behavior among recovering youth. Neurocognitive and psychiatric influences on adolescent drug treatment outcomes appear to be significant yet are poorly understood. Increasing our understanding of relationships between client characteristics, skill development during treatments, and subsequent outcomes should also help to improve adolescent drug treatments.

DETAILED DESCRIPTION:
This Stage II study is in response to NIDA's Behavioral Therapies Development Program (PA-99-107). A randomized clinical trial is proposed to evaluate the direct, mediated, and moderated effects of Integrated Family and Cognitive-Behavioral Therapy (IFCBT), a multisystems treatment for adolescent drug abuse with promising efficacy results. In the first study aim, we seek to evaluate the separate and possibly synergistic effects of family systems and cognitive-behavioral IFCBT components on posttreatment drug abuse problem severity, problem behavior, psychiatric distress, and academic achievement of adolescent drug abusers. Innovative analytic strategies are subsequently used to evaluate the degree to which successful outcomes are attributable to specific familial and cognitive-behavioral change processes targeted by IFCBT components. The possibility of effect-modification also is considered, with a focus on neurocognitive, psychiatric comorbidity, and demographic factors. Namely, we seek to understand how variations in specific client characteristics, such as executive dysfunctions or psychiatric comorbidity, might explain why treatments work for some drug abusing youths but not others. In addition to promising findings on IFCBT efficacy, this Stage II proposal benefits from the development and Stage I study application of (a) treatment manuals; (b) therapist training procedures; (c) therapist adherence and competence tools; (d) a neuropsychological battery to assess cognitive functions; (e) a psychodiagnostic battery to assess comorbid psychiatric disorders; and (f) a study assessment battery comprised of therapeutic process and outcome measures. This revised application has sought to address well-taken concerns cited by the reviewers while maintaining proposal strengths. The lack of adolescent drug treatment research continues to be a serious gap in the addictions literature despite alarmingly high rates of drug abuse among youth and the range of morbidities and mortality that result nationwide. If successful, this project should help to identify specific behavior change processes targeted by family systems and cognitive-behavioral treatments that foster subsequent reductions in drug use and problem behavior among recovering youth. Neurocognitive and psychiatric influences on adolescent drug treatment outcomes appear to be significant yet are poorly understood. Increasing our understanding of relationships between client characteristics, skill development during treatments, and subsequent outcomes should also help to improve adolescent drug treatments.

ELIGIBILITY:
Inclusion Criteria: Adolescents and young adults aged 13 to 21 years old who have significant drug-related problems or meet diagnostic criteria for drug abuse/dependence.

-

Exclusion Criteria: Acute psychotic, suicidal, homicidal ideation. Problem severity requiring residential treatment.

-

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2005-01; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Marijuana use abstinence and frequency | 3, 6, 9, 12, and 18 Month Follow-up Assessment
  The Personal Experience Inventory (PEI) is a youth self-report drug use inventory that assesses the frequency and quantity of substance use and drug abuse risk factors, such as deviant behavior and peer drug use.
Other drug use abstinence and frequency | 3, 6, 9, 12, 18 month Follow-up Assessment
  The Adolescent Stage of Change Scale (ASCS) consists of items to measure youths' motivation to change drug use behavior. Urine will also be analyzed for the presence of drugs, such as cannabinoids, cocaine, opiates, amphetamine, methamphetamine, MDMA, benzodiazepines, and barbiturates using gas chromatography/mass spectrometry methods.
Alcohol use abstinence and frequency | 3, 6, 9, 12, and 18 month Follow-up assement
  Personal Experience Inventory (PEI) is a youth self-report drug use inventory that assesses the frequency and quantity of substance use and drug abuse risk factors, such as deviant behavior and peer drug use.

SECONDARY OUTCOMES:
Legal involvement | 3,6,9, 12, and 18 month follow-up assessment
  The parent and adolescent versions of the Missouri Assessment for Genetics Interview for Children (MAGIC) address diagnostic symptoms associated with DSM-IV criteria including conduct disorder and antisocial personality disorder and includes questions on legal involvement.
Family functioning | 3,6,9,12, and 18 month follow-up assessment
  The Family Assessment Measure (FAM) is a self-report tool for parents and children that measures change processes targeted by the family systems component of IFCBT, including appropriate role performance, parental control, and communication.
Problem solving skill | 3,6,9,12, and 18 month assessment
  The Social Problem Solving Inventory (SPSI) assesses respondents' problem solving skill across the five dimensions addressed during the Problem Solving Therapy module of IFCBT.
Rational Beliefs | 3,6,9,12, and 18 month assessment
  The Rational Thinking Questionnaire assesses rational and irrational beliefs in relation to drug-related and general life issues.
Learning Strategy Skill | 3,6,9,12, and 18 month assessment
  The Motivated Strategies for Learning Questionnaire (MSLQ) assesses adolescents' motivation to learn in school and use of effective learning strategies that are addressed during the Learning Strategy Training module of IFCBT.
Academic Achievement | 3,6,9,12, and 18 month assessment
  The Interview on Sociodemographic Characteristics is administered to collect information on grades, academic achievement, days truant, school behavior problems, detention, suspension, and expulsion.

CONTACTS AND LOCATIONS:
Overall Officials: William W. Latimer, Ph.D., M.P.H., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Result] Latimer WW, Winters KC, D'Zurilla T, Nichols M. Integrated family and cognitive-behavioral therapy for adolescent substance abusers: a stage I efficacy study. Drug Alcohol Depend. 2003 Sep 10;71(3):303-17. doi: 10.1016/s0376-8716(03)00171-6. PMID 12957348
- [Result] Latimer WW, Stone AL, Voight A, Winters KC, August GJ. Gender differences in psychiatric comorbidity among adolescents with substance use disorders. Exp Clin Psychopharmacol. 2002 Aug;10(3):310-5. doi: 10.1037//1064-1297.10.3.310. PMID 12233992